CLINICAL TRIAL: NCT00891293
Title: A Second Open-Label Extension of a Double-Blind, Parallel, Phase IV Study to Assess the Efficacy and Safety of Adjunctive Lovaza® (Formerly Known as Omacor®) Therapy in Hypertriglyceridemic Subjects Treated With Antara™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111821
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Hypertriglyceridemia
Keywords: omega-3-acid ethyl esters; Very high triglycerides; Lovaza; fenofibrate
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fenofibrate; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) (Experimental): Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]
  Interventions: Drug: Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters)

INTERVENTIONS:
Drug: Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) — Open-label Antara (fenofibrate) + open-label Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]

SUMMARY:
This was a 24-month, open-label extension study that followed an 8-week double-blind study (Study LOV111859/OM5) and an 8-week, open-label extension study (LOV111860/OM5X). Study LOV111859/OM5 was conducted to evaluate whether combination therapy with Lovaza (omega-3-acid ethyl esters) and Antara (fenofibrate) would result in a greater reduction in serum triglyceride levels in hypertriglyceridemic subjects than treatment with fenofibrate alone. This second extension of 24 months was to assess the continued efficacy of adjunctive Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] therapy in hypertriglyceridemic subjects treated with Antara (fenofibrate) in lowering serum triglyceride (TG) levels.

DETAILED DESCRIPTION:
Three studies comprise this program. Study LOV111859/OM5 (double-blind study) was followed by two open label extensions - LOV111860/OM5X (1st open label extension - 8 weeks) and LOV111821/OM5XX (2nd open label extension - 24 months).

Studies LOV111859/OM5 and LOV111860/OM5X are outlined in NCT00246636.

ELIGIBILITY:
Subjects were men and women who had successfully completed the previous open-label extension study (LOV111860/OM5X) and had met all inclusion and exclusion criteria for the original double-blind study (LOV111859/OM5) and throughout LOV111860/OM5X, or who had a renewed waiver of a previously approved protocol deviation.

Eligibility for entry into this study was based on the inclusion/exclusion criteria described of the double-blind LOV111859/OM5 protocol.

Subjects were men and women who had successfully completed the previous open-label extension study (LOV111860/OM5X) and had met all inclusion and exclusion criteria for the original double-blind study (LOV111859/OM5) and throughout LOV111860/OM5X, or who had a renewed waiver of a previously approved protocol deviation. The main eligibility criteria for LOV111859/OM5 were,

* 18 to79 years of age (inclusive) at screening
* fasting serum TG levels ≥500 mg/dL and <1300 mg/dL
* BMI ≥ 25 kg/m2 and ≤43 kg/m2.

Subjects enrolled directly from the end of LOV111860/OM5X into LOV111821/OM5XX.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Duhwoody, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Bloomington, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Wentzville, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia

REFERENCES:
- [Background] Roth EM, Bays HE, Forker AD, Maki KC, Carter R, Doyle RT, Stein EA. Prescription omega-3 fatty acid as an adjunct to fenofibrate therapy in hypertriglyceridemic subjects. J Cardiovasc Pharmacol. 2009 Sep;54(3):196-203. doi: 10.1097/FJC.0b013e3181b0cf71. PMID 19597368

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovaza (Formerly Known as Omacor) and Fenofibrate: Open-label Lovaza (omega-3-acid ethyl esters)[formerly known as Omacor] 4 g/day and open-label fenofibrate 130 mg/day
Period: Overall Study
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Started | 93 (93 participants were enrolled; baseline data are provided for 89 participants (Safety Population).)
Completed | 9
Not Completed | 84
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 2
Not completed — Laboratory abnormality | 4
Not completed — Lost to Follow-up | 7
Not completed — Subject withdrew consent | 7
Not completed — Sponsor termination | 62

BASELINE CHARACTERISTICS:
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 52.4 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 69
Race/Ethnicity, Customized [Number; unit: participants]
  White | 81
  Hispanic or Latino | 2
  American Indian or Alaska Native | 1
  Asian | 3
  Black or African American | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Triglycerides From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension).
Description: Median Percent Change in Serum Triglycerides from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of Serum Triglycerides from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: Modified Intent-To-Treat (MITT) Population is defined as subjects who have a baseline assessment in Study LOV111859/OM5 and at least one on-therapy Study LOV111821/OM5XX efficacy assessment.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -60.6 (20.72) [-85.3 to 55.9]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -62.0 (32.33) [-88.9 to 115.0]
Statistical Analysis 1: Comparison: Lovaza (Formerly Known as Omacor) and Fenofibrate; For the MITT analysis, the method of last observation carried forward (LOCF) was applied. The LOCF is the value of a previous non-baseline visit (post-enrollment) carried forward to the subsequent visit, if missing; Test type: Superiority or Other; p = 0.9999, ANOVA; Median Difference (Net) = 3.3, 95% CI [-2.8 to 9.4], Standard Deviation 29.01 — Difference Between Percent Change from LOV111859/OM5 Baseline to LOV111860/OM5X End-of-Treatment and Percent Change from LOV111859/OM5 Baseline to LOV111821/OM5XX End-of-Treatment

2. Secondary Outcome: Percent Change in Total Cholesterol From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study).
Description: Median Percent Change in Total Cholesterol (Total-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of Total-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: MITT Population is defined as subjects who have a baseline assessment in Study LOV111859/OM5 and at least one on-therapy Study LOV111821/OM5XX efficacy assessment.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -6.7 [-47.6 to 25.3]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -13.2 [-55.1 to 20.1]

3. Secondary Outcome: Percent Change in VLDL-C From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study)
Description: Median Percent Change in very low density lipoprotein-cholesterol (VLDL-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of VLDL-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -58.3 [-82.2 to 14.9]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -54.6 [-88.4 to 10.5]

4. Secondary Outcome: Percent Change in LDL-C From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study)
Description: Median Percent Change in low density lipoprotein-cholesterol (LDL-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of LDL-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | 52.8 [-24.8 to 147.7]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | 37.5 [-49.0 to 159.7]

5. Secondary Outcome: Percent Change in HDL-C From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study)
Description: Median Percent Change in high density lipoprotein-cholesterol (HDL-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of HDL-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -3.0 [-62.9 to 44.1]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -11.1 [-47.2 to 175.6]

6. Secondary Outcome: Percent Change in Ratio of Total-C:HDL-C From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Ext. Study)
Description: Median Percent Change in the ratio of total cholesterol (Total-C) to high density lipoprotein-cholesterol (HDL-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change for the ratio of Total-C to HDL-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -4.8 [-45.2 to 234.6]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | 0 [-72.4 to 74.6]

7. Secondary Outcome: Percent Change in Apo A-1 From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study
Description: Median Percent Change in apolipoprotein (apo) A-1 from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of apo A-1 from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | 1.7 [-68.6 to 34.4]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | 2.9 [-20.4 to 179.1]

8. Secondary Outcome: Percent Change in Apo B From LOV111859/OM5 (Double-blind [DB[ Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study)
Description: Median Percent Change in apolipoprotein (apo) B from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of apo B from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | 0.0 [-39.9 to 47.6]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -7.3 [-59.3 to 35.4]

9. Secondary Outcome: Percent Change in Non-HDL-C From LOV111859/OM5 (Double-blind [DB] Study) Baseline to Week 8 of LOV111860/OM5X (1st Open-label [OL] Extension Study) and From LOV111859/OM5 (DB Study) Baseline to Month 24 of LOV111821/OM5XX (2nd OL Extension Study)
Description: Median Percent Change of non- high density lipoprotein-cholesterol (non-HDL-C) from the baseline of LOV111859/OM5 to the End-of-Treatment (EOT) (Week 8) of LOV111860/OM5X and Median Percent Change of non-HDL-C from the baseline of LOV111859/OM5 to the EOT (Month 24) of LOV111821/OM5XX.
Time Frame: LOV111859/OM5 Baseline to LOV111860/OM5X Week 8 and LOV111859/OM5 Baseline to LOV111821/OM5XX Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Number analyzed (Participants) | 89
Percentage change
  LOV111859/OM5 Baseline to LOV111860/OM5X EOT | -7.2 [-51.4 to 30.9]
  LOV111859/OM5 Baseline to LOV111821/OM5XX EOT | -13.3 [-64.8 to 20.1]

ADVERSE EVENTS:
Description: While 93 subjects were enrolled in the study, information for serious adverse events and other adverse events is provided for 89 subjects. These 89 subjects represent the Safety Population. The Safety Population is defined as all subjects who received a dose of study medication and had at least one post-enrollment safety assessment.
Arm/Group | Lovaza (Formerly Known as Omacor) and Fenofibrate
Serious Adverse Events (participants affected / at risk) | 4
Other Adverse Events (participants affected / at risk) | 47
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Lovaza (Formerly Known as Omacor) and Fenofibrate
Acute myocardial infarction (Cardiac disorders) | 1/89
Elevated liver function (Investigations) | 1/89
L2-3 herniated lumbar disk (Musculoskeletal and connective tissue disorders) | 1/89
R lower extremity cellulitus (Infections and infestations) | 1/89
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Lovaza (Formerly Known as Omacor) and Fenofibrate
Upper respiratory tract infection (Infections and infestations) | 15/89
Influenza (Infections and infestations) | 6/89
Hypertension (Vascular disorders) | 6/89
Back pain (Musculoskeletal and connective tissue disorders) | 5/89
Diabetes (Endocrine disorders) | 5/89
Sinusitis (Infections and infestations) | 5/89
Nausea (Gastrointestinal disorders) | 5/89

LIMITATIONS AND CAVEATS:
LOV111821/OM5XX was terminated due to the lack of substantial incremental change in the primary endpoint lipid values above that reached in either the original study (LOV111859/OM5) or the first extension study (LOV111860/OM5X).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.